CLINICAL TRIAL: NCT03146117
Title: Application of Integrated PET and Dual Energy CT Imaging for Staging and Imaged Based Radiotherapy Treatment Planning in Lung Cancer
Brief Title: PET-DECT for Staging and Imaged Based Radiotherapy Planning in Lung Cancer
Status: Terminated | Type: Observational
Why Stopped: Recruit completed
Sponsor: Medical University of South Carolina (Other)
Collaborators: Siemens Corporation, Corporate Technology (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00060975
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: PET CT
Keywords: PET CT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall goal of this project is to investigate the diagnostic performance of integrated F-18 fluorodeoxyglucose-positron emission tomography (FDG-PET) and Dual Energy CT (DECT) imaging in determining the thoracic nodal status of small-cell lung cancer (SCLC) and non-small-cell lung cancer (NSCLC), and its impact on target volume delineation for image guided radiation therapy (IGRT) planning.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study: (All answers must be "YES" for subject to be eligible.)

1. Subject must have a suspected SCLC or NSCLC.
2. Subject must be 18-90 years of age.
3. Subject must have been referred for a clinically indicated PET-CT.
4. Subject must provide written informed consent prior to any study-related procedures being performed.
5. Subject must be willing to comply with all clinical study procedures.

Exclusion Criteria:

The presence of the following excludes subjects from the study: (All answers must be "NO" for subject to be eligible.)

1. Subject is a pregnant or nursing female. Exclude the possibility of pregnancy:

   * By testing (serum or urine βHCG) within 24 hours before contrast agent administration, or
   * By surgical sterilization, or
   * Post-menopausal, with minimum one (1) year history without menses.
2. Subject has impaired renal function (eGFR<30 mL/min).
3. Subject has an acute psychiatric disorder or is cognitively impaired.
4. Subject is using or is dependent on substances of abuse.
5. Subject is unwilling to comply with the requirements of the protocol.
6. Subject has an allergy against iodinated contrast agents and cannot be premedicated.
7. Subject is in acute unstable condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators plan to recruit a total of 50 individuals (male, female; age range 18-90 years) referred to undergo a clinically indicated PET-CT examination. Patients will be identified from the Radiology department schedule. With the proposed 50 patient data set, the investigators are neither targeting nor avoiding the selective recruitment of women and minorities. Given the narrow inclusion criteria, the investigators plan to recruit patients irrespective of demographics. The patient will be approached by IRB-approved study personnel under the direction of one of the licensed physician investigators listed on the study, either prior to or on the day of the planned PET-CT examination (a single study visit, with the objective to perform the clinically indicated imaging), with a full explanation and request for consent as required by the IRB. MUSC policies regarding patient consent will be followed. The study design is not randomized.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
PET-CT accuracy for lung tumor and thoracic adenopathy detection | One year
  Knowledge gained during this study may potentially allow for an improvement in PET-CT accuracy for lung tumor and thoracic adenopathy detection, and for a more accurate definition of the RT target, decreasing the radiation dose delivered to normal tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo De Cecco, MD PHD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No